CLINICAL TRIAL: NCT05566821
Title: Scaling up Trauma and Violence-Informed Outreach With Women Affected by Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Inner-City Women's Initiatives Society (Unknown); Social Sciences and Humanities Research Council of Canada (Other); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Victoria Bungay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H22-01197
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gender-based Violence; Outreach Intervention
Keywords: Gender-based Violence; Trauma-informed; Outreach Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STRENGTH Outreach Intervention (Experimental): Participants enrolled in STRENGTH intervention elements
  Interventions: Behavioral: STRENGTH Outreach Intervention

INTERVENTIONS:
Behavioral: STRENGTH Outreach Intervention — The STRENGTH outreach intervention is a community-led, strengths-based, and trauma- and violence-informed program to support self-identifying women who experience interpersonal and structural gender-based violence. The outreach intervention aims to support individuals to achieve self-identified priorities.

SUMMARY:
Using a participatory action research design, this study examines the process and impact of implementing an evidence-informed, strengths-based, trauma- and violence-informed outreach program with women at greatest risk of health and social inequities to mitigate the effects of multiple forms of violence in their lives. Through collaboration among community service leaders and staff, women with lived or living experience of gender-based violence, and researchers, this project aims to improve the capacity of organizations to build and sustain effective and trusting relationships with women in order to foster health, well-being, safety, and increased ability to independently navigate their support needs.

DETAILED DESCRIPTION:
Using collaborative research activities, an advanced model of the STRENGTH intervention developed in earlier community-based studies is being tested. That evidence showed that women have unique strengths and abilities in navigating their safety, health and well-being, and that a strengths-based approach is critical to communicate respect and build trusting relationships. Trust facilitates women's engagement and retention in health and social care and enhances their capacities to independently navigate these systems. Appropriate, safe, and responsive outreach can effectively improve safety, reduce overdose deaths, and enhance engagement with health and social care.

The study involves a case-based mixed method design to test an empirically driven model for outreach with women affected by violence, through a series of longitudinal studies with diverse sub-groups of women in differing social and geographical contexts. The two-year intervention study is embedded in a larger 7-year national project aimed at building capacity of outreach programs to prevent and mitigate the effects of gender-based violence and advance the theory and practice of community-based, participatory action research.

Intervention-specific Research Questions:

1. How effective is this outreach program in:

   * building trusting relationships with women?
   * supporting women to achieve their self-identified priorities and goals (short-term, medium-term, and long-term goals) in ways that foster safety, autonomy and rights to self-determination?
2. What factors enable or confound the success of the outreach intervention?

Project Objectives

To generate new knowledge about program delivery to effectively engage with women to:

* Build trusting relationships between women and short-term, medium-term and long-term supports
* Enhance women's capacity for autonomy, ability and confidence in achieving short-, medium-, and long-term goals
* To generate new knowledge about how to enhance delivery of health and social care services that are non-harmful and non-traumatizing

This research will provide important knowledge about how to more effectively design, implement and evaluate programs and practices that can increase social and health supports and mitigate the effects of gender-based and structural violence. It tests how an empirically driven model of outreach combined with enhanced service integration supports women to identify their priority needs and can bridge the gap in service needs and access with women affected by violence and inequities.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a woman, therefore the study is trans-inclusive
* Have some degree of English proficiency in understanding and communication
* Live and/or spend significant time for work and/or health and social services in the service area of one of the participating community organizations
* Age 18 or over

Exclusion Criteria:

* Individuals not meeting the inclusion criteria listed above will be excluded from participation.
* In addition, women already enrolled in another program with wrap-around supports and who are able to independently navigate health and social care will not be eligible to participate in the outreach program intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identifying women
Enrollment: 39 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in trust from baseline to 3 months | Baseline (6 weeks post-enrollment) & 3 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 3 months post-baseline
Change in trust from baseline to 6 months | Baseline (6 weeks post-enrollment) & 6 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 6 months post-baseline
Change in trust from baseline to 9 months | Baseline (6 weeks post-enrollment) & 9 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 9 months post-baseline
Change in trust from baseline to 12 months | Baseline (6 weeks post-enrollment) & 12 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 12 months post-baseline
Safety in Care Encounters at Baseline | Baseline (6 weeks post-enrollment)
  Self-reported safety in clinical care encounters over the past three months using rating of 1 to 5 with higher scores being higher safety
Safety in Care Encounters at 3 months | 3 months post-baseline
  Self-reported safety in clinical care encounters over the past three months using rating of 1 to 5 with higher scores being higher safety
Safety in Care Encounters at 6 months | 6 months post-baseline
  Self-reported safety in clinical care encounters over the past three months using rating of 1 to 5 with higher scores being higher safety
Safety in Care Encounters at 9 months | 9 months post-baseline
  Self-reported safety in clinical care encounters over the past three months using rating of 1 to 5 with higher scores being higher safety
Safety in Care Encounters at 12 months | 12 months post-baseline
  Self-reported safety in clinical care encounters over the past three months using rating of 1 to 5 with higher scores being higher safety
Safety in Home Setting at Baseline | Baseline (6-weeks post-enrollment)
  Self-reported safety in current home setting for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Home Setting at 3 months | 3 months post-baseline
  Self-reported safety in current home setting for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Home Setting at 6 months | 6 months post-baseline
  Self-reported safety in current home setting for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Home Setting at 9 months | 9 months post-baseline
  Self-reported safety in current home setting for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Home Setting at 12 months | 12 months post-baseline
  Self-reported safety in current home setting for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Community Setting at Baseline | Baseline (6-weeks post-enrollment)
  Self-reported safety in community for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Community Setting at 3 months | 3 months post-baseline
  Self-reported safety in community for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Community Setting at 6 months | 6 months post-baseline
  Self-reported safety in community for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Community Setting at 9 months | 9 months post-baseline
  Self-reported safety in community for the previous three months using a rating of 1 to 5 with higher scores being higher safety
Safety in Community Setting at 12 months | 12 months post-baseline
  Self-reported safety in community for the previous three months using a rating of 1 to 5 with higher scores being higher safety

SECONDARY OUTCOMES:
Priorities achieved at 3 months | 3 months
  Were participants' self-identified priorities achieved after 3 months of intervention (yes/no)
Priorities achieved at 6 months | 6 months
  Were participants' self-identified priorities achieved after 6 months of intervention (yes/no)
Priorities achieved at 9 months | 9 months
  Were participants' self-identified priorities achieved after 9 months of intervention (yes/no)
Priorities achieved at 12 months | 12 months
  Were participants' self-identified priorities achieved after 12 months of intervention (yes/no)
Priorities achieved at 15 months | 15 months
  Were participants' self-identified priorities achieved after 15 months of intervention (yes/no)
Priorities achieved at 18 months | 18 months
  Were participants' self-identified priorities achieved after 18 months of intervention (yes/no)
Priorities achieved at 21 months | 21 months
  Were participants' self-identified priorities achieved after 21 months of intervention (yes/no)
Priorities achieved at 24 months | 24 months
  Were participants' self-identified priorities achieved after 24 months of intervention (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Bungay, PhD, Principal Investigator — Professor
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No